CLINICAL TRIAL: NCT02598427
Title: Phase I Dose Escalation Trial of Intrathecal Pertuzumab and Trastuzumab in Patients With New Untreated Asymptomatic or Low Symptomatic Brain Metastasis
Brief Title: Intrathecal Pertuzumab and Trastuzumab in Patients With New Untreated Asymptomatic or Low Symptomatic Brain Metastasis in HER2 Positive Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Inadequate enrollment
Sponsor: Kimberly Blackwell (Other)
Responsible Party: Sponsor-Investigator, Kimberly Blackwell, Professor of Medicine, Director of the Duke Breast Cancer Program, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00061309
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: HER2 Positive Untreated Metastatic Breast Cancer; Asymptomatic or Low Symptomatic Brain Metastasis in Breast Cancer
Keywords: Breast Cancer; HER2 Positive; HER2+; Brain Metastases; Metastatic Breast Cancer; Intrathecal Treatment; Lumbar Puncture; Pertuzumab; Trastuzumab; Advanced Breast Cancer; Duke University
MeSH Terms: conditions — Breast Neoplasms; Brain Neoplasms | interventions — pertuzumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intrathecal Pertuzumab and Trastuzumab (Experimental): Four cohorts will enroll in a dose escalation of pertuzumab and a consistent dose of trastuzumab. The cohorts will be assigned as follows:
  Cohort: Intrathecal Dose:
  1. 10mg pertuzumab, 80mg trastuzumab
  2. 20mg pertuzumab, 80mg trastuzumab
  3. 40mg pertuzumab, 80mg trastuzumab
  4. 80mg pertuzumab, 80mg trastuzumab
  Interventions: Drug: Pertuzumab; Drug: Trastuzumab

INTERVENTIONS:
Drug: Pertuzumab — Pertuzumab will be administered intrathecally via a lumber puncture. The dosing cohorts are described above in the arm description.
  Other Names: Perjeta
Drug: Trastuzumab — Trastuzumab will be administered intrathecally via a lumber puncture. The dosing cohorts are described above in the arm description.
  Other Names: Herceptin

SUMMARY:
The purpose of this research study is to determine how well pertuzumab and trastuzumab works in treating breast cancer that has spread to the brain. Pertuzumab and trastuzumab are treatments that stop breast cancer cells from growing abnormally by inhibiting (or blocking) members of a family of proteins that include Human Epidermal Growth Factor Receptor 2 (HER2).

Pertuzumab and trastuzumab have been found to be very effective for HER2-positive breast cancer and are FDA approved for treatment of metastatic breast cancer outside of the brain when given through the vein. This suggests that pertuzumab and trastuzumab may help shrink or stabilize HER2-positive breast cancer that has spread to the brain in this research study.

In this research study, the investigators are looking to see whether pertuzumab and trastuzumab will work to decrease the size of or stabilize breast cancer that has spread to the brain.

DETAILED DESCRIPTION:
Intrathecal administration of pertuzumab and trastuzumab will occur via lumbar puncture (spinal tap) under fluoroscopic guidance by interventional radiology at Duke University Medical Center. The spinal needle will be inserted into the spinal column and 7 mL of cerebrospinal fluid (CSF) will be collected. Once the CSF is removed, the intrathecal pertuzumab and trastuzumab will be administered using aseptic technique. At certain time points the CSF will be analyzed for free cell DNA. If subjects consent, the CSF fluid will also be stored for additional future research.

Patients will be treated using a 3+3 dose-escalation design. Patients will not be accrued to the next cohort (dose escalation) until at least one patient on the previous cohort has been followed for six weeks. If a dose limiting toxicity (DLT) is seen in a patient then the cohort will be expanded by an additional 3 patients to allow for 1 in 6 patients per cohort to have a DLT before dose escalation. Dose limiting toxicity will be assessed weekly during the first six weeks of the treatment.

Patients will be treated weekly for the first six weeks and then every 3 weeks (q21 days). Once the maximum tolerated dose is reached, an additional 12 patients will be enrolled in the cohort at the maximum tolerated dose. The maximum number of enrolled patients is 36. Dosing is as follows: Cohort 1 - 80mg IT trastuzumab, 10mg IT pertuzumab, cohort 2 - 80mg IT trastuzumab, 20mg IT pertuzumab, cohort 3 - 80mg IT trastuzumab, 40mg IT pertuzumab, cohort 4 - 80mg IT trastuzumab, 80mg IT pertuzumab. If the lowest dose level is found to be too toxic, the trial will stop without finding a maximum tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

* HER2 positive by 2013 ASCO-CAP guidelines (IHC 3+ and/or FISH positive; IHC 2+ HER2 patients are eligible with reflex FISH positive testing with the ratio ≥ 2.0) breast cancer patients with untreated asymptomatic or minimally symptomatic brain metastasis by MRI. There is no upper or lower limit to the size or number of brain metastases.
* Patients can have previous brain metastasis that was completely surgically resected if the previously resected lesion is at least 1 cm from target lesion(s) for this study. The location of the previous resection cavity is determined by the post-resection MRI.
* Patients can have previous brain metastasis that was treated with stereotactic radiosurgery (SRS) if the previously treated lesion is at least 1cm from the target lesion(s) for this study. The location of the previous SRS treatment location is determined by the SRS MRI.
* Patients can be on steroids as long as the dose has been stable for ≥ 7 days
* No limitations on prior systemic or intrathecal therapies.
* There are no restrictions on systemic therapy at enrollment.
* Negative serum pregnancy test for pre-menopausal women and women within 12 months from the onset of menopause.
* Sexually active women of childbearing potential must commit to 2 methods of contraception while enrolled on the trial and continue using contraceptives for at least 7 months post study drug administration. Sexually active men must commit to 1 method of contraception while enrolled and for 7 months after. Hormonal contraceptives such as birth control pills, patches, implants or injections are not allowed in patients who are HR+.
* Life expectancy ≥ 8 weeks
* Laboratory criteria: normal renal function: creatinine < 1.5 x upper limit of normal (ULN)), liver function: bilirubin ≤ 1.5 x ULN, transaminases ≤ 2 x ULN, except in known hepatic disease, wherein may be ≤ 5 x ULN, and blood counts: WBC ≥ 2.0, Neutrophils ≥1500, platelets ≥100,000, Hemoglobin ≥ 10.
* LVEF (left ventricular ejection fraction) ≥ 50%
* Karnofsky performance status (KPS) ≥ 50
* Age ≥ 18 years
* Patients must have the ability to give informed consent.
* Patients must sign an informed consent form.

Exclusion Criteria:

* No seizures, focal weakness of any extremity (by neurologic exam), or stroke symptoms in the past month.
* No history of prior whole brain radiation.
* No history of lumbar surgery or other pre-existing spinal conditions that would preclude frequent, safe, reliable lumbar punctures.
* No history of serious cardiac arrhythmia or EF < 50%.
* Systemic sites of disease need to be stable on systemic therapy based on the most recent (within 12 weeks) staging scans.
* Radiation while on study is not allowed EXCEPT to a localized region for pain control.
* No history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix) unless the patient has been in remission and off all other cancer therapy for at least 3 years.
* Patients should have no significant psychiatric illness or medical illness that would preclude the ability to comply with the protocol.
* Patients may not be pregnant or breastfeeding.
* No known hypersensitivity to trastuzumab or pertuzumab.
* Symptomatic intrinsic lung disease or extensive tumor involvement in the lungs resulting in dyspnea at rest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-02-22 (Actual); Study Completion 2018-02-22 (Actual)

PRIMARY OUTCOMES:
Safety as measured by adverse events | Baseline up to 36 weeks
  Adverse events will be closely monitored and assessed for all subjects on study treatment. The main observational portion of study will be complete at 36 weeks. However, subjects will be allowed to continue on treatment for as long as they are receiving clinical benefit and any adverse events occurring during this time will be assessed. Following discontinuation of study treatment, patient follow-up will take place every 3 months.
Maximum tolerated dose as measure by dose limiting toxicity | Baseline up to 36 weeks
  Toxicity will be graded according to the NCI-CTC version 4 and will be assessed weekly for the first six weeks of treatment and then every 21 days. A DLT is defined as any grade 3 or higher non-hematologic toxicity or grade 4 hematologic toxicity that occurs within the first 6 weeks of treatment that is assessed as possibly related to the intrathecal therapy. Any treatment delays occurring during the first six weeks of treatment that are due to study treatment-related toxicity will also be considered a DLT.
  The main portion of study will be complete at 36 weeks. However, subjects will be allowed to continue on treatment for as long as they are receiving clinical benefit.

SECONDARY OUTCOMES:
Response rate as measured by brain MRI | Every 6 weeks from Baseline up to 36 weeks
  Response assessed:
  Complete Response (CR): Radiographic complete response (RCR), 100% reduction in tumor, with complete clearing of MRI scan evidence of disease on 2 consecutive scans 6 weeks apart with stable or improved clinical function.
  Partial Response (PR): Radiographic stability of disease (RSD), > 50% but < 100% reduction in tumor, with improved clinical function.
  Stable Disease (SD): Radiographic stability of disease (RSD), < 50% reduction in tumor or < 25% increase in size of tumor, with stable clinical function.
  Progressive Disease (PD): Radiographic progressive disease (RPD), > 25% increase in size of tumor, and/or the presence of declining clinical function attributable to the CNS metastasis. Other indications of progression include development of new CNS metastases or increase in size of previous CNS metastasis. Changes in size of previous CNS metastasis must measure > 25% increase in the largest unidimensional measurement in the absence of new neurologic symptoms.
Changes in cell-free circulating tumor DNA (ctDNA) in response to treatment | Baseline up to 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Blackwell, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States